CLINICAL TRIAL: NCT01834378
Title: Diabetes Prevention in Primary Health Care With Special Emphasis on Physical Activity.
Brief Title: Diabetes Prevention in Clinical Practice.
Acronym: DIAVIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAVIP-1204; Swedish Research Council (Other Grant/Funding Number: Swedish Research Council)
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; insulin resistance; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Motor Activity

ARMS (3):
- No intervention (No Intervention)
- Low intensity intervention (Experimental)
  Interventions: Behavioral: Low intensity intervention
- High intensity intervention (Experimental)
  Interventions: Behavioral: High intensity intervention.

INTERVENTIONS:
Behavioral: Low intensity intervention — We administer, a pedometer and the participants receive a prescription on physical exercise.
  Arms: Low intensity intervention
Behavioral: High intensity intervention. — We schedule group sessions for changes in behavior e.g. type of physical activity to prefer, barriers for change of life style etc.
  Arms: High intensity intervention

SUMMARY:
We randomize individuals with impaired glucose tolerance to one of three arms for degree of physical activity: 1. Continue with your current life style; 2. Ordinary life activities for increased physical activity; 3. Scheduled group activities for changed behavior. The overall aim is to focus on change of physical activity and to keep other life style activities more or less unchanged (diet, smoking, etc) and the effect on metabolic variables.

ELIGIBILITY:
Inclusion Criteria:

1. Impaired glucose tolerance
2. Age: 20-85yrs

Exclusion Criteria:

1. Type2 diabetes
2. Significant disease making life style changes unlikely to happen
3. Unable to communicate in Swedish

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
HOMA IR | 12 months after inclusion (baseline)
  Insulin resistance according to HOMA